CLINICAL TRIAL: NCT01981460
Title: PhotoDynamic Therapy for Line Infection Prevention (PLIP): Pilot Study on Normal Volunteers
Brief Title: PhotoDynamic Therapy for Line Infection Prevention (PLIP): Pilot Study on Healthy Volunteers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeanine Wiener-Kronish, Chief of Anesthesia, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P-002692
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Light; Therapy, Complications
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroprep and biopatch (No Intervention): Both arms are cleaned with chloroprep and a biopatch is placed on each arm.
- Methylene blue and light treatment (Experimental): Methylene blue and light treatment for 17 minutes are done twice over 1 week intervals.
  Interventions: Procedure: Methylene blue and light treatment

INTERVENTIONS:
Procedure: Methylene blue and light treatment — Methylene blue and light treatment for 17 minutes are done twice over 1 week intervals.
  Arms: Methylene blue and light treatment

SUMMARY:
We are evaluating the effect of methylene blue and visible light activation on the microbiome of the skin.

DETAILED DESCRIPTION:
Antiseptics are routinely utilized to prevent infections of vascular catheters. We are evaluating the addition of methylene blue and light activation on skin to determine whether this inexpensive and non-toxic treatment can decrease skin pathogens and prevent blood stream infections of long-term vascular catheters. This is a pilot study of normal volunteers to determine the effect on the microbiome of the addition of methylene blue and light activation on antiseptic-treated skin.

ELIGIBILITY:
Inclusion Criteria:

* Normal individuals without skin problems

Exclusion Criteria:

* Smokers
* Diabetics
* Atopic dermatitis
* G-6-PD deficiency
* Eczema
* Other skin conditions
* Allergies to methylene blue or chlorhexadine

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the skin microbiome after methylene blue treatment | 1 week
  We compared the two arms of each subject --one arm treated with chloraprep and a biopatch [routine treatment of skin] to the routine treatment with the addition of methylene blue spray and light activation. The microbiome of both skin areas were assessed before and after the routine treatment and the treatment with the addition of methylene blue therapy;

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine Wiener-Kronish, MD, Principal Investigator — MGH